CLINICAL TRIAL: NCT01446276
Title: Long-term Investigation of Resveratrol on Lipid Turnover in Obese Men With Nonalcoholic Fatty Liver Disease. Effects on Liver Fat Content and Basal and Insulin Stimulated FFA and VLDL-triglyceride Metabolism
Brief Title: Long-term Investigation of Resveratrol on Fat Metabolism in Obese Men With Nonalcoholic Fatty Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: The Ministry of Science, Technology and Innovation, Denmark (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: M-20110172A
Record Dates: First submitted 2011-10-03; First posted 2011-10-05 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2013-10

CONDITIONS: Obesity; Nonalcoholic Fatty Liver Disease
Keywords: Obesity; Resveratrol; Nonalcoholic fatty liver disease; Insulin sensitivity; Lipid turnover; Liver fat content
MeSH Terms: conditions — Obesity; Non-alcoholic Fatty Liver Disease; Insulin Resistance | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Resveratrol (Experimental): Resveratrol 500mg 3 times daily for six month
  Interventions: Dietary Supplement: Resveratrol
- Placebo (Placebo Comparator): Placebo 1 tablet 3 times daily for six month
  Interventions: Other: Placebo
- Control group (No Intervention): Men without non-alcoholic fatty liver disease

INTERVENTIONS:
Dietary Supplement: Resveratrol — 500 mg 3 times daily for six month
  Arms: Resveratrol
Other: Placebo — 1 placebo tablet 3 times daily for six month
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate potential metabolic effects of resveratrol in obese healthy men with non-alcoholic fatty liver disease.

The investigators hypothesize that resveratrol will:

* decrease hepatic very-low-density-lipoprotein-triglyceride (VLDL-TG) secretion
* decrease liver fat content
* increase insulin sensitivity

The investigators will look at changes in:

* lipid turnover (VLDL-TG kinetics, palmitate kinetics, indirect calorimetry)
* liver fat content (MR liver spectroscopy)
* insulin sensitivity (glucose kinetics during hyperinsulinaemic euglycaemic clamp)
* body composition (DXA and MRI)
* lipase activity and fat cell size (fat biopsy from abdominal and femoral adipose tissue)

ELIGIBILITY:
Inclusion Criteria:

* Male
* 25-65 years
* Obesity (BMI > 28 kg/m2, waist/hip ratio > 0,95)
* Have nonalcoholic fatty liver disease (NAFLD)(intervention group) or do not have NAFLD (control group)
* May have hypertension and/or hypercholesterolemia
* Written informed consent

Exclusion Criteria:

* Any other disease than NAFLD (e.g. diabetes, thyroid or parathyroid disease, heart, liver or kidney disease)
* Present and previous malignancy
* Alcohol dependency (more than 21 units of alcohol per week)
* History of smoking
* Participation in studies with radioactive isotopes within the last six months
* Hemoglobin under normal range regarding to sex (under 8.3 mmol/l for men)

Ages: 25 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Hepatic VLDL-TG secretion and peripheral VLDL-TG clearance | six month
  - Changes from baseline after treatment with either resveratrol or placebo

SECONDARY OUTCOMES:
Basal and insulin stimulated free fatty acid (FFA) and glucose turnover | six month
  - Changes from baseline after treatment with either resveratrol or placebo
VLDL-TG oxidation | six month
  - Changes from baseline after treatment with either resveratrol or placebo
Body composition (fat mass, fat-free mass, percent fat, visceral fat mass) | six month
  - Changes from baseline after treatment with either resveratrol or placebo
lipoprotein lipase activity and fat cell size in abdominal and femoral adipose tissue biopsy | six months
  - Changes from baseline after treatment with either resveratrol or placebo
Baseline data | Baseline
  - Comparison of baseline data between intervention group and control group

CONTACTS AND LOCATIONS:
Overall Officials: Søren Nielsen, MD, associate professor, DMSc, Study Chair — Department of Endocrinology and Internal Medicine
Locations (1):
- Department of Endocrinology and Internal Medicine, Aarhus C, Denmark

REFERENCES:
- [Derived] Poulsen MK, Nellemann B, Bibby BM, Stodkilde-Jorgensen H, Pedersen SB, Gronbaek H, Nielsen S. No effect of resveratrol on VLDL-TG kinetics and insulin sensitivity in obese men with nonalcoholic fatty liver disease. Diabetes Obes Metab. 2018 Oct;20(10):2504-2509. doi: 10.1111/dom.13409. Epub 2018 Jul 5. PMID 29885082
- [Derived] Poulsen MK, Nellemann B, Stodkilde-Jorgensen H, Pedersen SB, Gronbaek H, Nielsen S. Impaired Insulin Suppression of VLDL-Triglyceride Kinetics in Nonalcoholic Fatty Liver Disease. J Clin Endocrinol Metab. 2016 Apr;101(4):1637-46. doi: 10.1210/jc.2015-3476. Epub 2016 Feb 1. PMID 26829441